CLINICAL TRIAL: NCT07030634
Title: Effect of Adding Blood Flow Restriction and Proprioception Training to Traditional Rehabilitation on Ankle Joint Sensations
Brief Title: Blood Flow Restriction and Proprioception Training on Ankle Joint Sensations
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed fekry ibrahim salman, assistant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BFR and proprioception
Record Dates: First submitted 2025-06-03; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Lateral Ankle Sprain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group (A) (Active Comparator): A (control group) received conventional physical therapy only
  Interventions: Other: conventional physical therapy
- Group (B) (Experimental): Experimental Group B received conventional physical therapy with Low load blood flow restriction
  Interventions: Other: conventional physical therapy; Other: Low load blood flow restriction
- Group (C) (Experimental): received conventional physical therapy with proprioception training
  Interventions: Other: conventional physical therapy; Other: proprioception training
- Group (D) (Experimental): received conventional physical therapy, Low load blood flow restriction and proprioception training.
  Interventions: Other: conventional physical therapy; Other: Low load blood flow restriction; Other: proprioception training

INTERVENTIONS:
Other: conventional physical therapy — consist of Strengthening exercise: will begin with isometric exercises performed against an immovable object in four directions of ankle movement (dorsiflexion, planter flexion, inversion, and eversion) and will be progressed to dynamic resistive exercises (isotonic exercises) using ankle weights.
  and Bracing: The participants will receive instructions from the therapist about using and applying the soft brace. The soft brace will be based on the principles of the functional tape bandage
Other: Low load blood flow restriction — Patients in blood flow restriction training groups will receive low load resistance exercise (20-40 % 1RM) using tourniquet around thigh proximally to knee joint to occlude arterial blood flow by 50-80 %.
  Arms: Group (B); Group (D)
Other: proprioception training — Patients will receive proprioception exercises in duration of 30 minutes per session, frequencies will be 3 times per week, and lengths for 4 weeks (Matthew et al., 2017). Progression of the proprioceptive training should be static to dynamic (such as lateral movements, backward movements, jumping, cutting, twisting, pivoting), slow speeds to faster speeds with balance and control, two legs to one leg, and with visual control to no visual control.
  Arms: Group (C); Group (D)

SUMMARY:
Thirty-four participants with grade I and II recurrent ankle sprain, were referred from orthopaedic physician. Their ages ranged from 20 to 30 years old. All participants will be divided randomly into two groups A, B. Seventeen participants per group. Participant selected from both sexes, with body mass index between 18 and 24.9 Kg/m², with self-reported history of at least one significant lateral ankle sprain (LAS) greater than 12 months prior to testing and recurring ankle sprains, ankle "giving way" and/or "feelings of instability". Participants with previous surgery or fracture and with any adverse effects to blood occlusion will be excluded.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be selected from both sexes.
* Participants BMI will be between 18 and 24.9 (Kg/m²).
* Dominant or non-dominant lower limb .
* Grade I, and II recurrent ankle sprain patients .
* Participants self-reported a history of at least one significant lateral ankle sprain (LAS) greater than 12 months prior to testing, and recurring ankle sprains, ankle "giving way," and/or "feelings of instability."
* Participant will have unilateral recurrent ankle sprain

Exclusion Criteria:

* A history of previous surgeries to the musculoskeletal structures (ie, bones, joint structures, nerves) in either limb of the lower extremity.
* A history of a fracture in either limb of the lower extremity requiring realignment .
* Acute injury to musculoskeletal structures of other joints of the lower extremity in the previous 3 months, which impacted joint integrity and function (ie, sprains, fractures) resulting in interruption of desired physical activity .
* Hip joint or, Knee joint replacement .
* Patients possibly at risk of adverse reactions of blood flow restriction are those with poor circulatory system, obesity, diabetes, arterial calcification, sickle cell trait, severe hypertension, or renal compromise
* Any neurological conditions which affect proprioception such as polyneuropathy, multiple sclerosis, and sensory ataxia .
* Vestibular deficits, and vision problems .
* Pregnancy.

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-20 (Estimated)

PRIMARY OUTCOMES:
peak torque of ankle muscles | after three times weekly physiotherapy sessions for four consecutive weeks.
  Each participant will be seated on the dynamometer chair in a relaxed position with the hip joint slightly flexed and the knee flexed about 45° so that the fulcrum of the dynamometer will be corresponded to the axis of the participant's ankle joint with the foot resting on the ankle attachment in a neutral position between dorsi flexion and planter flexion; standard toe straps will be used over the foot. Also, two straps will be wrapped around theextremity proximal to the patella and the pelvis to minimize movements of the trunk, hip, and knee during testing, which would interfere with the ankle measurement
limits of stability | after three times weekly physiotherapy sessions for four consecutive weeks.
  Before the start of each testing session, the Biodex will be calibrated according to the manufacturer's manual. The participants will be familiarized with testing procedures through free practical sessions to minimize the learning effects that occur during testing. All measurements will be performed at level eight of stability (the most suitable level), and the test duration will be set at 20 seconds for three successive trials. Each participant will be tested for stability index (SI) and limits of stability (LOS). The limits of stability (LOS) are defined as the area that the subject safely moves without changing the base of support. The stability index (SI) represents the patient's ability to control balance and motor control skills at 50% LOS

IPD SHARING:
Plan to Share IPD: Undecided